CLINICAL TRIAL: NCT04517903
Title: Validation Study on Eye Rubbing Questionnaire in Patients With or Suspected of Having a Keratoconus (KC)
Acronym: QFK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2019/53
Record Dates: First submitted 2020-08-14; First posted 2020-08-19 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Keratoconus
Keywords: Keratoconus; Eye rubbing
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Intervention Model Description: eye rubbing questionnaire at baseline and 15 days later
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- exploratory phase (Experimental): eye rubbing questionnaire at baseline and 15 days later
  Interventions: Other: eye rubbing questionnaire

INTERVENTIONS:
Other: eye rubbing questionnaire — eye rubbing questionnaire at baseline and 15 days later for exploratory phase; at baseline and then validation by a Group Nominal

SUMMARY:
KC is a degenerative disorder of the cornea. Keratoconus etiopathogenesis remains unclear and may rely on environmental and genetic factors. Usually considered as a rare disease (<1/2000), but the prevalence is nowadays growing worldwide up to 1/500. In that pathology, cornea progressively gets thinner, and there is a deformation of the corneal surface which can induce high order optical aberrations and visual impairment.

Eye rubbing is certainly the main factor in the progression or development of keratoconus (KC), yet it is only very partially evaluated and quantified in current management. Environmental and clinical factors will be collected and associated with a eye rubbing Questionnaire, specifically pointing out eye rubbing.

DETAILED DESCRIPTION:
CNRK center is working on an eye rubbing questionnaire since 2017 in order to quantify that pejorative factor. Patient education can limit in a certain amount the Keratoconus progression. Thus, our objective will be to evaluate the therapeutic impact on Keratoconus progression of patient's education against eye rubbing according to an eye rubbing Questionnaire.

The validation of a dedicated questionnaire is an important act that will allow the scientific evaluation of this factor with both environmental and behavioral traits. It can thus be integrated into our care activity for its intrinsic educational and therapeutic virtues and for its decision-making aid for certain treatments. It will be useful first of all for the refinement of the correct prescription of corneal collagen crosslinking for evolving KC or KC with a high risk of progression.

ELIGIBILITY:
Inclusion Criteria:

* Coming for the first time for expert advice on KC
* Having a suspected or known KC
* Being over 13 years old (or from 13 years old)
* Possess computer connection equipment (computer, tablet or smartphone) and access to the network, for the completion of the questionnaire at home.
* Being affiliated to or beneficiary of health insurance
* Have signed the informed consent form from the patient and from legal representatives for minor patient

Exclusion Criteria:

* Being incapacitated or unable to follow study procedures
* Patient under legal protection
* Previous ocular surgery

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
validation of our eye rubbing questionnaire | Baseline and 15 days after (Day 15)
  validation of our eye rubbing questionnaire will be made through the evaluation of its Suitability (Appearance validity, Content validity), Reliability (Consistency and homogeneity, Reproducibility), Applicability (Feasibility and acceptability), Validity (Construct validity), Sensitivity (Sensitivity to change, Discriminative validity)

SECONDARY OUTCOMES:
questionnaire simplification | Month 6
  Statistical criteria for questionnaire simplification: ceiling and floor effects, response rates, correlations, reproducibility, measurement error and internal consistency. These elements are part of the content validity and reliability stages of the COSMIN recommendations
Expert consensus by nominal group | Month 6
  Expert consensus by nominal group. This is the only method suitable for validating a clinical questionnaire

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - CHU Bordeaux, Bordeaux
  - CHU Brest, Brest
  - CHU de Clermont-Ferrad, Clermont-Ferrand
  - Hospices Civils de Lyon, Lyon
  - CHU de Montpellier, Montpellier
  - Centre National Ophtalmologique des Quinze Vingt, Paris
  - CHU de Rouen, Rouen
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No